CLINICAL TRIAL: NCT01594892
Title: Dose-intensified Image-Guided Fractionated Radiosurgery for Spinal Metastases (DOSIS)
Brief Title: Fractionated Radiosurgery for Painful Spinal Metastases
Acronym: DOSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOSIS
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Neoplasm Metastasis; Neoplastic Processes; Neoplasm Recurrence, Local; Neoplasm, Residual; Pain
Keywords: Spinal metastases; Vertebral metastases; Radiosurgery; Radiotherapy; Stereotactic body radiotherapy; Pain
MeSH Terms: conditions — Neoplasm Metastasis; Neoplastic Processes; Neoplasm Recurrence, Local; Neoplasm, Residual; Pain | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Evaluation of the single intervention - dose-intensified SBRT
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose intensified SBRT (Experimental): Depending on the modified Mizumoto Score (0-4 points or 5-9 points) patients will be treated with 10 fractions of 4.85Gy in involved parts of the vertebra and 3Gy in not-involved parts using a simultaneous integrated boost or with 5 fractions of 7Gy in involved parts of the vertebra and 4Gy in not-involved parts using a simultaneous integrated boost, respectively.
  Interventions: Radiation: Radiosurgery

INTERVENTIONS:
Radiation: Radiosurgery — Fractionated radiosurgery using intensity-modulated treatment planning and volumetric image-guided treatment delivery

SUMMARY:
It is the study hypothesis that hypo-fractionated image-guided radiosurgery significantly improves pain relief compared to historic data of conventionally fractionated radiotherapy. Primary endpoint is pain response 3 months after radiosurgery, which is defined as pain reduction of ≥2 points at the treated vertebral site on the 0 to 10 Visual Analogue Scale. 60 patients will be included into this II trial.

DETAILED DESCRIPTION:
The current study will investigate efficacy and safety of radiosurgery for painful vertebral metastases and three characteristics will distinguish this study.

1. A prognostic score for overall survival will be used for selection of patients with longer life expectancy to allow for analysis of long-term efficacy and safety.
2. Fractionated radiosurgery will be performed with the number of treatment fractions adjusted to either good (10 fractions) or intermediate (5 fractions) life expectancy. Fractionation will allow inclusion of tumors immediately abutting the spinal cord due to higher biological effective doses at the tumor - spinal cord interface compared to single fraction treatment.
3. Dose intensification will be performed in the involved parts of the vertebrae only, while uninvolved parts are treated with conventional doses using the simultaneous integrated boost concept.

ELIGIBILITY:
Inclusion Criteria:

1. Established histological diagnosis of a malignant tumour (primary or metastatic)
2. Vertebral metastasis confirmed via biopsy or radiology
3. Pain in the involved spinal region or free of pain under pain medication
4. Fully consenting patients, >18 years old
5. Karnofsky Performance Index ≥60%
6. Good or intermediate life expectancy according to the modified prognostic Mizumoto Score (score ≤ 9)
7. Patient must be able to tolerate fixation systems and 30 minutes treatment time
8. Discussed in interdisciplinary tumour board
9. The following types of spinal tumours are eligible:

   * Recurrent / residual tumours after surgery
   * Tumours in medically inoperable patients or patients deemed inoperable due to limited life expectancy / tumour load
   * Lesions associated with significant surgical risk

Exclusion Criteria:

1. Short life expectancy according to the modified Mizumoto Sore
2. "Radiosensitive" histologies (i.e. lymphoma, SCLC, multiple myeloma)
3. Non-ambulatory status
4. Progressive neurological symptoms/deficit
5. > 3 involved vertebral levels
6. > 2 treatment sites
7. Spine instability
8. Previous radiotherapy at the involved levels

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2015-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of patients, in whom pain is decreased in response to treatment | Change in pain from baseline to 3 months post-treatment
  Decrease in pain by ≥2 points at the treated vertebral site on the 0 (no pain) to 10 (the severest pain) Visual Analogue Scale without analgesic increase

SECONDARY OUTCOMES:
Local tumor control | 2 years
  At the treated vertebral levels assessed with MRI
Local tumor control | 2 years
  At the treated vertebral levels assessed with CT imaging
Overall survival | 2 years
  Death from any cause
Patient-assessed 5 dimensions of patient's quality-of-life | Changes in quality of life from baseline to 3 months post-treatment
  Measured with the 5-level (no problems, slight problems, moderate problems, severe problems, and extreme problems) EuroQol 5-Dimension Questionnaire (EQ-5D) questionnaire
Patient-assessed overall health status | Changes in quality of life from baseline to 3 months post-treatment
  Measured with the EuroQol Visual Analog Scale from 0 ("the worst health you can imagine") to 100 (the best health you can imagine")
Number of patients developing acute toxicity | Changes from baseline up to 6 weeks post-treatment
  Measured with NCI CTCAE v 4.0
Number of patients developing late toxicity | Changes from >6weeks up to 2 years post-treatment
  Measured with NCI CTCAE v 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, MD, Principal Investigator — Department of Radiation Oncology, University of Wuerzburg
Locations (5):
- Germany (2):
  - Leopoldina Schweinfurt, Schweinfurt
  - Department of Radiation Oncology, University of Wuerzburg, Würzburg
- Netherlands Cancer Institute, Amsterdam, Netherlands
- University Hospital Zurich, Zurich, Switzerland
- The Royal Marsden Hospital NHS Foundation Trust, Sutton, United Kingdom

REFERENCES:
- [Background] Guckenberger M, Hawkins M, Flentje M, Sweeney RA. Fractionated radiosurgery for painful spinal metastases: DOSIS - a phase II trial. BMC Cancer. 2012 Nov 19;12:530. doi: 10.1186/1471-2407-12-530. PMID 23164174
- [Result] Guckenberger M, Sweeney RA, Hawkins M, Belderbos J, Andratschke N, Ahmed M, Madani I, Mantel F, Steigerwald S, Flentje M. Dose-intensified hypofractionated stereotactic body radiation therapy for painful spinal metastases: Results of a phase 2 study. Cancer. 2018 May 1;124(9):2001-2009. doi: 10.1002/cncr.31294. Epub 2018 Mar 2. PMID 29499073
- [Derived] Mantel F, Sweeney RA, Klement RJ, Hawkins MA, Belderbos J, Ahmed M, Toussaint A, Polat B, Flentje M, Guckenberger M. Risk factors for vertebral compression fracture after spine stereotactic body radiation therapy: Long-term results of a prospective phase 2 study. Radiother Oncol. 2019 Dec;141:62-66. doi: 10.1016/j.radonc.2019.08.026. Epub 2019 Sep 13. PMID 31526672